CLINICAL TRIAL: NCT03132428
Title: Multicenter, Prospectively Defined Observational Registry With Retrospective Data Collection, Evaluating Premature and Term-Near-Term Neonates With Pulmonary Hypertension Receiving Inhaled Nitric Oxide Via Invasive or Noninvasive Ventilation
Brief Title: Registry to Evaluate INOmax in Newborn Babies With Pulmonary Hypertension
Acronym: PaTTerN
Status: Terminated | Type: Observational
Why Stopped: Positive results at interim analysis
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Other Study IDs: MNK19050056
Record Dates: First submitted 2017-04-25; First posted 2017-04-27 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Pulmonary Hypertension of Newborn
Keywords: Premature and term-near-term neonates
MeSH Terms: conditions — Premature Birth | interventions — Endothelium-Dependent Relaxing Factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- P Neonates: Premature (P) neonates [at least 27 weeks but less than 34 weeks of gestational age]
  Interventions: Drug: INOmax
- TNT Neonates: Term-Near-Term (TNT) neonates at least 34 weeks of gestational age
  Interventions: Drug: INOmax

INTERVENTIONS:
Drug: INOmax — Nitric oxide gas for inhalation provided via mechanical ventilation or non invasive ventilation

SUMMARY:
Pulmonary hypertension is high blood pressure in the arteries to the lungs. It is a serious condition. It causes the blood vessels that carry blood from the heart to the lungs to become hard and narrow. When this happens, the heart has to work harder to pump the blood through.

Some babies are born with pulmonary hypertension (PH). Doctors might use INOmax (a gas the baby breathes) to help newborn babies (neonates) with PH. This study will use information from the records of registered babies to see how effective and safe INOmax is for treating premature and other newborn babies for up to 11 days after they are born.

ELIGIBILITY:
Inclusion Criteria:

1. Was either a P neonate born at least 27 weeks to less than 34 weeks of gestational age (GA) or a TNT neonate born at least 34 weeks but no more than 40 weeks of GA.
2. Was administered INOmax therapy after birth to 7 days of age via any route (invasive or noninvasive ventilation) for a minimum treatment period of at least 24 hours up to 96 ± 12 hours. The participants may receive INOmax for a longer period.
3. Had PH, as confirmed by echocardiogram or a differential saturation gradient of at least 10%.
4. Received INOmax administration as part of routine clinical practice in a Level III or higher neonatal intensive care unit in the United States.
5. Has all variables required to calculate OI or SOI (a baseline sample prior to treatment and 4 samples obtained during treatment).

Exclusion Criteria:

1. Was at risk of imminent death (death expected within 24 hours).
2. Received extracorporeal membrane oxygenation (ECMO).
3. Had a life-threatening abnormality (cranial, cardiac, thoracic), chromosomal abnormality, congenital diaphragmatic hernia, congenital heart defect (other than patent ductus arteriosus or small atrial septal defect).
4. Had been resuscitated requiring chest compressions within 6 hours of receiving INOmax.
5. Had Grade IV bilateral intraventricular hemorrhage or periventricular leukomalacia.
6. Had active uncontrolled bleeding.
7. Had disseminated intravascular coagulopathy.
8. Had active seizures while receiving anticonvulsants.
9. Experienced prolonged asphyxia with evidence of severe acidosis (pH < 7.25).
10. Received concomitant pulmonary vasodilator therapy (eg, prostacyclin or sildenafil) except when sildenafil was used to wean the participant from INOmax therapy.

Ages: 27 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature (P) and term-near-term (TNT) neonates
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
Number of neonates with significant response to INOmax treatment within each age group | within 108 hours
  Significant response is defined as at least a 25% improvement from baseline in oxygenation index or surrogate oxygenation index (OI/SOI) during INOMAX treatment

SECONDARY OUTCOMES:
Number of neonates with significant response to Inomax treatment within each age group and severity group | within 108 hours
  The severity of pulmonary hypertension (PH) is classified for each participant Categories: Mild, Moderate, Severe
Time to reach significant response to Inomax treatment within each age group and severity group | within 108 hours
  The median time to INOmax complete response (25% improvement) for neonates with each baseline PH severity classification Categories: Mild, Moderate, Severe
Number of neonates with partial response to INOmax treatment within each age group and severity group | within 108 hours
  Partial response is defined as less than a 25% improvement in OI/SOI during INOmax treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Leader, Study Director — Mallinckrodt
Locations (30):
- United States (30):
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - Loma Linda University Health Care, Loma Linda, California
  - Miller Children's and Women's Hospital - Long Beach, Long Beach, California
  - Children's Hospital of Orange County, Orange, California
  - Sharp Mary Birch Hospital for Women and Newborns, San Diego, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Yale New Haven Children's Hospital, New Haven, Connecticut
  - Florida Hospital for Children, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - University of Chicago Comer Children's Hospital, Chicago, Illinois
  - University of Iowa Stead Family Children's Hospital, Iowa City, Iowa
  - University of Kentucky Chandler, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - University of Minnesota Amplatz Children's Hospital, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Saint Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of New Jersey at Newark Beth Israel Medical Center, Newark, New Jersey
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Hospital at OU Medical Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nelin L, Kinsella JP, Courtney SE, Pallotto EK, Tarau E, Potenziano JL. Use of inhaled nitric oxide in preterm vs term/near-term neonates with pulmonary hypertension: results of the PaTTerN registry study. J Perinatol. 2022 Jan;42(1):14-18. doi: 10.1038/s41372-021-01252-x. Epub 2021 Oct 28. PMID 34711938